CLINICAL TRIAL: NCT05964088
Title: Mortality and Morbidity Associated With New Onset Acute Kidney Injury in Critically Ill COVID-19 Infection Patients
Status: Completed | Type: Observational
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Principal Investigator, Michael Neeki, Attending Physician, Arrowhead Regional Medical Center
Other Study IDs: 22-18
Record Dates: First submitted 2023-07-24; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1: These critically ill patients were directly admitted to the intensive care unit from the emergency department
- Group 2: These critically ill patients were were initially managed on the medical floor and later transferred to the intensive care unit for worsening respiratory status

SUMMARY:
This study explored the incidence of morbidity and mortality associated with AKI in critically ill adult patients infected with COVID-19. There are two groups for comparison. Group1. patients were directly admitted to the intensive care unit (ICU) from the emergency department (ED) Group 2. patients were initially managed on the medical floor and later transferred to the ICU for worsening respiratory status. The investigating team evaluated the correlation of inflammatory markers and common risk factors such as obesity, diabetes, hypertension and ethnicity to the development of AKI in the target population. The primary outcome is mortality participants will received their regular healthcare in a medical setting

ELIGIBILITY:
Inclusion Criteria:

positive for SARS-CoV-2 on a real-time polymerase chain reaction test (RT-PCR) upon admission to the hospital

Exclusion Criteria:

chronic kidney disease end stage renal disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a two-year retrospective study of critically ill adult patients infected with COVID-19 that were admitted to the intensive care unit on ventilatory support. Patients included in this study were admitted to Arrowhead Regional Medical Center (ARMC) from March 1, 2020 to February 12, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Mortality | from admission until death from any cause, whichever comes first, assessed up to three months
  mortality at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Neeki, DO, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

REFERENCES:
- [Derived] Fischer N, Miao X, Weck D, Matalon J, Neeki CC, Pennington T, Dong F, Arabian S, Neeki MM. Mortality and morbidity associated with new onset acute kidney injury in critically ill COVID-19 infection patients. Int J Emerg Med. 2024 Jul 29;17(1):97. doi: 10.1186/s12245-024-00666-6. PMID 39075369